CLINICAL TRIAL: NCT05040477
Title: Comparison of Muscle Energy Technique and Facet Joint Mobilization in the Patient With Chronic Neck Pain.
Brief Title: Muscle Energy Technique and Facet Joint Mobilization in Chronic Neck Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00868 Huma Tabassum
Record Dates: First submitted 2021-08-05; First posted 2021-09-10 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Chronic Neck Pain
Keywords: cervical pain; chronic neck pain,; Muscle energy technique,; Facet join mobilization,; cervical lordosis,; cervical curve
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group (1): Muscle energy techniques,Moist Hot pack and TENS. (Experimental): Experimental group included Moist Hot pack of 14/15' over cervical region for 15 mins. Hydro collator Temperature according to standardized hot pack is 40-45C.Conventional TENS applied for 10 mins.
  Baseline NPRS, NDI, Cervical ROMs, and posterior tangent angle.These pre and post intervention values were mentioned in questionnaire. The participants were administered with muscle energy technique (PIR) and data was collected again 2 and 4 weeks after the interventions.
  Interventions: Other: Muscle energy Technique
- Experimental Group (2): Facets joint mobilizations, Moist Hot pack and TENS. (Experimental): Experimental group includedMoist Hot pack of 14/15' over cervical region for 15 mins. Hydro collator Temperature according to standardized hot pack is 40-45οC.Conventional TENS applied for 10 mins.
  Baseline NPRS, NDI, Cervical ROMs, and posterior tangent angle. These pre and post intervention values were mentioned in questionnaire. The participants were administered with Facet joint mobilization (UPA & SNAGS) and data was collected again 2 and 4 weeks after the interventions.
  Interventions: Other: Muscle energy Technique
- Control Group:Conventional Therapy (Stretching, strengthening , Moist Hot pack and TENS) (Active Comparator): Control group includedMoist Hot pack of 14/15' over cervical region for 15 mins. Hydro collator Temperature according to standardized hot pack is 40-45οC.Conventional TENS applied for 10 mins.
  Baseline NPRS, NDI, Cervical ROMs, and posterior tangent angle. These pre and post intervention values were mentioned in questionnaire. The participants were administered with Conventional (sustained stretching and isometric strengthening) physical therapy and data was collected again 2 and 4 weeks after the interventions.
  Interventions: Other: Muscle energy Technique

INTERVENTIONS:
Other: Muscle energy Technique — Muscle Energy technique was used to increase the strength of weak muscles,relaxation of tightened muscles in result mobilizes the restricted joint segments.MET's group received 3-5 repetition of post isometric relaxation (PIR).
  Treatment through Facet Joint Mobilization based on 3 sets of 15 repetitions of unilateral poster-anterior glide (UPA) using initially grade I & II mobilizations followed by grade III of mitland glides on selected tender segments and 5 repetitions of extension sustained natural apophyseal glides (SNAGs) on hypo mobile segments.
  Conventional therapy comprising of stretching and isometric strengthening exercises in combination with TENS and heat therapy.
  Other Names: Facet Joint Mobilization; Conventional Therapy

SUMMARY:
The purpose of the study is to compare the muscle energy technique, facet joint mobilization and conventional physical therapy in individuals with chronic neck pain on cervical lordosis, cervical range of motions, numeric pain rating scale and NDI. A randomized control trial was conducted at physiotherapy department of HIT hospital, Taxila Cantt. The sample size was 105 calculated through open-epi tool. The participants were divided into three interventional groups, experimental group (1), experimental group (2), and control group (3) each having 35 participants. The study duration was six months. Sampling technique applied was Purposive sampling for recruitment and group randomization using sealed envelope method. Only 35 to 50 years participants with 4-8 pain intensity on NPRS in cervical region were included in the study. Goniometer, Posterior tangent method on lateral radiographs for cervical curve and Self structured Questionnaire. Data was collected at baseline then 2 and 4 weeks after the application of interventions. Data analyzed through SPSS version 21.

ELIGIBILITY:
Inclusion Criteria:

* Chronic patients (more than 12 weeks)
* Male and female patients
* Patients having recurrence of neck pain at least once in the last month.
* Patients from the age group of 35-50 years.
* Patients having mechanical neck pain ranging from 4-8 on Numeric Pain Rating Scale (NPRS).
* Cervical straightening on X-rays.
* Limited &painful cervical Rang of motion (ROMs)

Exclusion Criteria:

* Any recent history of trauma, active inflammation, Tumor, vertebra-basilar insufficiency and cervical myelopathy & radiculopathy.
* No history of serious underlying pathology, nerve root compromise, structural changes and deformities, genetic spinal disorders or previous spinal surgery

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2020-08-30 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Cervical Lordosis Measurement (posterior tangent method) | 4 week
  measure cervical lordosis by drawing tangent line along posterior border of C2 to C7 vertebra and measuring posterior tangent angle on lateral radio graph of cervical spine.At baseline and 4 weeks after baseline
Numeric pain rating scale | 4 week
  Will utilize for measurement of neck pain intensity.Minimum pain score is labeled as "zero" and maximum pain score is labeled as "10".At baseline, 2 and 4 weeks after baseline.

SECONDARY OUTCOMES:
Neck disability index: | 4 week
  Will utilize for measurement of functional disability level among patients with chronic neck pain.At baseline, 2 and 4 weeks after baseline
Cervical goniometry: | 4 week
  Will utilize to measure range of motions for all movement at cervical spine with the help of valid & reliable tool, goniometer.At baseline, 2 and 4 weeks after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Lal Gul Khan, MS, Principal Investigator — Riphah International University
Locations (1):
- HIT Taxila Cantt Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borisut S, Vongsirinavarat M, Vachalathiti R, Sakulsriprasert P. Effects of strength and endurance training of superficial and deep neck muscles on muscle activities and pain levels of females with chronic neck pain. J Phys Ther Sci. 2013 Sep;25(9):1157-62. doi: 10.1589/jpts.25.1157. Epub 2013 Oct 20. PMID 24259936
- [Background] Akhter S, Khan M, Ali SS, Soomro RR. Role of manual therapy with exercise regime versus exercise regime alone in the management of non-specific chronic neck pain. Pak J Pharm Sci. 2014 Nov;27(6 Suppl):2125-8. PMID 25410083
- [Background] 3. Gautam R, Dhamija JK, Puri A, Trivedi P, Sathiyavani D, Nambi G. Comparison of Maitland and Mulligan mobilization in improving neck pain, ROM and disability. Int J Physiother Res. 2014;2(3):561-6.
- [Background] Andersen LL, Saervoll CA, Mortensen OS, Poulsen OM, Hannerz H, Zebis MK. Effectiveness of small daily amounts of progressive resistance training for frequent neck/shoulder pain: randomised controlled trial. Pain. 2011 Feb;152(2):440-446. doi: 10.1016/j.pain.2010.11.016. Epub 2010 Dec 21. PMID 21177034
- [Background] 5. Sutjana IDP, Erg M, PFK S, Erg A, Sutjana IDP, Irfan M, et al. Pemberian Teknik Mulligan Dan Soft Tissue Mobilization Lebih Baik Daripada Hanya Soft Tissue Mobilization Dalam Meningkatkan Lingkup Gerak Sendi Ekstensi, Rotasi, Lateral Fleksi Cervical Pada Mechanical Neck Pain. Sport and Fitness Journal. 2013;1(2).
- [Background] Yoon SY, Moon HI, Lee SC, Eun NL, Kim YW. Association between cervical lordotic curvature and cervical muscle cross-sectional area in patients with loss of cervical lordosis. Clin Anat. 2018 Jul;31(5):710-715. doi: 10.1002/ca.23074. Epub 2018 Apr 14. PMID 29575212
- [Background] Scheer JK, Tang JA, Smith JS, Acosta FL Jr, Protopsaltis TS, Blondel B, Bess S, Shaffrey CI, Deviren V, Lafage V, Schwab F, Ames CP; International Spine Study Group. Cervical spine alignment, sagittal deformity, and clinical implications: a review. J Neurosurg Spine. 2013 Aug;19(2):141-59. doi: 10.3171/2013.4.SPINE12838. Epub 2013 Jun 14. PMID 23768023
- [Background] Page P. Current concepts in muscle stretching for exercise and rehabilitation. Int J Sports Phys Ther. 2012 Feb;7(1):109-19. PMID 22319684
- [Background] 9. Chaitow L, Crenshaw K. Muscle energy techniques: Elsevier Health Sciences; 2006
- [Background] 10. Kage V, Bootwala F, Kudchadkar G. Effect of Bowen Technique versus Muscle Energy Technique on Asymptomatic Subjects with Hamstring Tightness: A Randomized Clinical Trial. International Journal of Medical Research & Health Sciences. 2017;6(4):102-8.
- [Background] Peng B, Pang X, Li D, Yang H. Cervical spondylosis and hypertension: a clinical study of 2 cases. Medicine (Baltimore). 2015 Mar;94(10):e618. doi: 10.1097/MD.0000000000000618. PMID 25761188
- [Background] Buyukturan O, Buyukturan B, Sas S, Kararti C, Ceylan I. The Effect of Mulligan Mobilization Technique in Older Adults with Neck Pain: A Randomized Controlled, Double-Blind Study. Pain Res Manag. 2018 May 15;2018:2856375. doi: 10.1155/2018/2856375. eCollection 2018. PMID 29861800
- [Background] 13. Hing W, Hall T, Rivett DA, Vicenzino B, Mulligan B. The Mulligan Concept of Manual Therapy-eBook: Textbook of Techniques: Elsevier Health Sciences; 2015.
- [Background] 14. Maitland G, Bank K. Vertebral manipulation 2002. Butterworth Heinemann, Oxford
- [Background] Osama M, Tassadaq N, Malik RJ. Effect of muscle energy techniques and facet joint mobilization on spinal curvature in patients with mechanical neck pain: A pilot study. J Pak Med Assoc. 2020 Feb;70(2):344-347. doi: 10.5455/JPMA.14189. PMID 32063632
- [Background] 16. Gupta S, Jaiswal P, Chhabra D. A comparative study between postisometric relaxation and isometric exercises in non-specific neck pain. Journal of exercise science and physiotherapy. 2008;4(2):88-94.
- [Background] 17. Sharma A, Angusamy R, Kalra S, Singh S. Efficacy of post-isometric relaxation versus integrated neuromuscular ischaemic technique in the treatment of upper trapezius trigger points. Indian Journal of Physiotherapy and Occupational Therapy. 2010;4(3):1-5.
- [Background] 18. Sharmila B. Isometric muscle energy technique and non-specific neck pain in secondary school teachers-results of an experimental study. Indian Journal of Physiotherapy and Occupational Therapy. 2014;8(2):58.
- [Background] 19. Mahajan R, Kataria C, Bansal K. Comparative effectiveness of muscle energy technique and static stretching for treatment of subacute mechanical neck pain. Int J Health Rehabil Sci. 2012;1(1):16-21.
- [Background] 20. Rana AA, Ahmad A, Gillani SA, Idrees MQ, Awan I. Effects of conventional physical therapy with and without muscle energy techniques for treatment of Upper Cross Syndrome. Rawal Medical Journal. 2020;45(1):127-32
- [Background] 21. Pragassame SA, Kurup VM, Kour J. Efficacy of sustained natural apophyseal glides mulligan technique on mobility and function in patients with cervical spondylosis: An experimental study. Journal of Natural Science, Biology and Medicine. 2020;11(2):128
- [Background] 22. Al Shehri A, Khan S, Shamsi S, Almureef SS. COMPARATIVE STUDY OF MULLIGAN (SNAGS) AND MAITLAND MOBILIZATION IN NECK PAIN. European Journal of Physical Education and Sport Science. 2018
- [Derived] Tabassum H, Mariam M, Gondal KS. Comparison of muscle energy technique and facet joint mobilisation in the patient with chronic neck pain: A randomized controlled trial. J Pak Med Assoc. 2024 Jan;74(1):10-15. doi: 10.47391/JPMA.9206. PMID 38219157